CLINICAL TRIAL: NCT05426265
Title: The Effects of Videogames on Depression Symptoms and Brain Dynamics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aalto University (Other)
Collaborators: Business Finland (Other); Helsinki University Central Hospital (Other); Turku University Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MelioraRCT
Record Dates: First submitted 2022-05-17; First posted 2022-06-21 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Major Depressive Disorder
Keywords: Depression; Digital therapeutics; Digital mental health intervention
MeSH Terms: conditions — Depressive Disorder, Major; Depression

STUDY DESIGN:
Intervention Model Description: The effectiveness of MEL-T01 and comparator MEL-S01 are studied. Their effectiveness is compared to a treatment-as-usual (TAU) group who also receive the intervention after a 12 week waiting period.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The research design is randomized and double-blinded. Subject randomization in study arms as well as treatment is automatized.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- MEL-T01 (Experimental): MEL-T01 is a game-based digital-therapeutics (DTx) medical software device that implements personalised cognitive training to alleviate MDD symptoms and improve cognitive performance in MDD subjects.
  Interventions: Device: MEL-T01
- MEL-S01 (Active Comparator): MEL-S01 is an active comparator similar to MEL-T01 but without personalized cognitive training elements.
  Interventions: Device: MEL-S01
- TAU (No Intervention): Treatment-as-usual.

INTERVENTIONS:
Device: MEL-T01 — A 12 week intervention with MEL-T01.
  Other Names: Meliora
  Arms: MEL-T01
Device: MEL-S01 — A 12 week intervention with MEL-S01.
  Arms: MEL-S01

SUMMARY:
The purpose of the study is to evaluate the effects of a game-based digital-therapeutics (DTx) medical software device on the symptoms of depression in adults with confirmed major depressive disorder.

DETAILED DESCRIPTION:
The study is a comparator-controlled, randomised, double-blinded intervention study aimed at assessing the effects of the investigational device MEL-T01, "Meliora", on the symptoms of major depressive disorder (MDD). MEL-S01 acts as a comparator. MEL-T01 is a game-based digital-therapeutics (DTx) medical software device developed at Aalto University and is intended to be used as a treatment for MDD together with treatment-as-usual (TAU). MEL-T01 implements personalised cognitive training to alleviate MDD symptoms and improve cognitive performance in MDD subjects.

Subjects volunteering to participate in this investigation are adults whose MDD is confirmed through MINI interview. They have an on-going mental health treatment contact with a mental health professional. The subjects are randomised into three arms with equal probabilities in blocks of six consecutive subjects. Subjects in the MEL-T01 and MEL-S01 arms are engaged in the intervention for 12 weeks while those in the TAU arm are on a follow-up period during these 12 weeks. After this 12-week period, the subjects in MEL-T01 and MEL-S01 arms enter a 12-week follow-up period and the subjects in TAU arm engage with either the MEL-T01 or MEL-S01 intervention (randomised at T0 with equal probability) for 12 weeks.

The subjects are recommended to play the investigational-device game for a total of 48 hours during the 12 weeks of active intervention with a recommended weekly dose of 4 hours. A minimum of 24 hours is needed for inclusion to hypothesis testing. The subjects are limited to a daily maximum of 1.5 hours of game time.

The subjects' mental health symptoms and well-being are evaluated through online questionnaires five times: before subjects are randomised into one of the three groups (T0), and then 4 (T1), 8 (T2), 12 (T3), and 24 (T4) weeks after the study has begun.

ELIGIBILITY:
Inclusion Criteria:

* Between 18-65 year-old
* Suffering from major depressive disorder
* Have an ongoing mental health treatment contact to basic healthcare, specialised healthcare, student healthcare or occupational healthcare
* Has sufficient eyesight with or without prescription
* Has a Windows computer with internet connection and mouse
* Has email and phone number

Exclusion Criteria:

* They have threat of self-harm
* They have addiction to digital games
* They have psychotic disorders
* They are pregnant or breastfeeding
* They have impaired ability in decision making
* They are prisoner or forensic subject
* They have neurological disorders such as epilepsy or brain injury

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1001 (Actual)
Dates: Start 2022-06-28 (Actual); Primary Completion 2024-08-14 (Actual); Study Completion 2024-08-14 (Actual)

PRIMARY OUTCOMES:
PHQ-9 total change from baseline to posttreatment: experimental group vs. treatment as usual group | Day 0 to Day 84
  The patient health questionnaire (PHQ-9, Kroenke et al., 2001) is a self-report measure of major depressive disorder. The PHQ-9 scores each of the nine DSM-IV criteria for MDD from "0" (not at all) to "3" (nearly every day), providing a 0-27 severity score of depression. The higher the total score the more severe the depression.
  The change in the PHQ-9 total score between before the 12 week intervention and after the intervention is measured. The change score of MEL-T01 group is compared with the change score of the treatment-as-usual (TAU) group.
PHQ-9 total change from baseline to posttreatment: active comparator group vs. treatment as usual group | Day 0 to Day 84
  The patient health questionnaire (PHQ-9, Kroenke et al., 2001) is a self-report measure of major depressive disorder. The PHQ-9 scores each of the nine DSM-IV criteria for MDD from "0" (not at all) to "3" (nearly every day), providing a 0-27 severity score of depression. The higher the total score the more severe the depression.
  The change in the PHQ-9 total score between before the 12 week intervention and after the intervention is measured. The change score of MEL-S01 group is compared with the change score of the treatment-as-usual (TAU) group.
PHQ-9 total change from baseline to posttreatment: experimental group vs. active comparator group | Day 0 to Day 84
  The patient health questionnaire (PHQ-9, Kroenke et al., 2001) is a self-report measure of major depressive disorder. The PHQ-9 scores each of the nine DSM-IV criteria for MDD from "0" (not at all) to "3" (nearly every day), providing a 0-27 severity score of depression. The higher the total score the more severe the depression.
  The change in the PHQ-9 total score between before the 12 week intervention and after the intervention is measured. The change score of MEL-T01 group is compared with the change score in the MEL-S01 group.

SECONDARY OUTCOMES:
QIDS total change from baseline to posttreatment | Day 0 to Day 84
  The quick inventory of depressive symptomatology (QIDS-SR16) is a self-report measure comprising of 16 questions on a scale of 0-3 which assess the severity of depressive symptoms. The inventory provides a total score between 0 and 48: the higher the total score the more severe the depression.
  For each of the three study arms, the change in total QIDS-SR16 scores between before the intervention and after the 12 week intervention is measured. Then, the average change scores in each of the three groups are compared with each other.
RRS (short version) total change from baseline to posttreatment | Day 0 to Day 84
  Ruminative Response Scale (RRS), short version, is an eight item self-report questionnaire that uses a four point Likert-scale. This leads to a total score between 8 and 64 where higher values indicate higher depressive brooding.
  For each of the three study arms, the change in total RRS scores between before the intervention compared and after the 12 week intervention are measured. Then, the average change scores in each of the three groups are compared with each other.
GAD-7 total change from baseline to posttreatment | Day 0 to Day 84
  The general anxiety disorder scale (GAD-7) is a seven-item self-report questionnaire that uses a 4-point scale (between 0 and 3) to evaluate the degree of anxiety symptoms. The questionnaire provides a total between 0 and 21: the higher the total score, the more severe the anxiety.
  For each of the three study arms, the change in total GAD-7 scores between before the intervention and after the 12 week intervention is measured. Then, the average change scores in each of the three groups are compared with each other.
SDS total change from baseline to posttreatment | Day 0 to Day 84
  The Sheehan disability scale (SDS) is a self-administered three item questionnaire using a 11-point scale (between 0 and 10). The scale is used to measure functional impairment. The scale provides a total score between 0 and 30: the higher the score, the higher the functional impairment. In addition, the scale measures "the number of days lost to symptoms" and "the number of days unproductive due to the symptoms".
  For each of the three study arms, the change in total SDS scores between before the intervention and after the 12 week intervention is measured. Then, the average change scores in each of the three groups are compared with each other.
PVSS total change from baseline to posttreatment | Day 0 to Day 84
  The positive valence systems scale (PVSS) is a 21-item self-report questionnaire using a scale from 1 to 9. This leads to a total score between 21 and 189 where a lower total score indicates higher anhedonia.
  For each of the three study arms, the change in total PVSS scores between before the intervention and after the 12 week intervention is measured. Then, the average change scores in each of the three groups are compared with each other.
WHO-5 total change from baseline to posttreatment | Day 0 to Day 84
  The well-being index (WHO-5) is a five item self-report questionnaire using a scale from 0 to 5. This leads to a total score is between 0 and 25: higher scores indicate higher subjective well-being.
  For each of the three study arms, the change in total WHO-5 scores between before the intervention and after the 12 week intervention is measured. Then, the average change scores in each of the three groups are compared with each other.
Correlation between PHQ-9 total change and playing time in group MEL-T01 | Day 0 to Day 84
  The patient health questionnaire (PHQ-9, Kroenke et al., 2001) is a self-report measure of major depressive disorder. The PHQ-9 scores each of the nine DSM-IV criteria for MDD from "0" (not at all) to "3" (nearly every day), providing a 0-27 severity score of depression. The higher the total score the more severe the depression.
  For the treatment MEL-T01 group, the change scores in the total PHQ-9 score between before the intervention and after the 12 week intervention is measured. Then, the correlation between the change score and the minutes played during the intervention is calculated. This leads to a correlation score that evaluates whether a higher symptom change is associated with higher playing time.
Correlation between PHQ-9 total change and playing time in group MEL-S01 | Day 0 to Day 84
  The patient health questionnaire (PHQ-9, Kroenke et al., 2001) is a self-report measure of major depressive disorder. The PHQ-9 scores each of the nine DSM-IV criteria for MDD from "0" (not at all) to "3" (nearly every day), providing a 0-27 severity score of depression. The higher the total score the more severe the depression.
  For the active comparator MEL-S01 group, the change scores in the total PHQ-9 score between before the intervention and after the 12 week intervention is measured. Then, the correlation between the change score and the minutes played during the intervention is calculated. This leads to a correlation score that evaluates whether a higher symptom change is associated with higher playing time.
Correlation between PHQ-9 total change and IEQ in group MEL-T01 | Day 0 to Day 84
  The immersive experiences questionnaire (IEQ, Jennett et al., 2008) is a self-report questionnaire that measures the subjective experience of being immersed while playing a video game. It has 31 questions on a scale of 1-7. This creates a total score between 31 and 217: the higher totals indicate higher immersion. In addition, there is one question - "How immersed did you feel?" - on a scale of 1-10.
  For the treatment MEL-T01 group, we measure the correlation between 1) the change in the total PHQ-9 score between before the intervention and after the 12 week intervention and 2) the total IEQ score (excluding the one additional questionnaire) as measured after the 12 week intervention.
  This leads to a correlation score that evaluates whether a higher symptom change is associated with higher immersion in the game.
Correlation between PHQ-9 total change and IEQ in group MEL-S01 | Day 0 to Day 84
  The immersive experiences questionnaire (IEQ, Jennett et al., 2008) is a self-report questionnaire that measures the subjective experience of being immersed while playing a video game. It has 31 questions on a scale of 1-7. This creates a total score between 31 and 217: the higher totals indicate higher immersion. In addition, there is one question - "How immersed did you feel?" - on a scale of 1-10.
  For the treatment MEL-S01 group, we measure the correlation between 1) the change in the total PHQ-9 score between before the intervention and after the 12 week intervention and 2) the total IEQ score (excluding the one additional questionnaire) as measured after the 12 week intervention.
  This leads to a correlation score that evaluates whether a higher symptom change is associated with higher immersion in the game.

OTHER OUTCOMES:
GAS total change from baseline to posttreatment | Day 0 to Day 84
  The game addiction scale (GAS, Lemmens et al., 2009) is a self-report 7-item questionnaire using a 1-5 scale which measures game addiction. This provides a total between 7 and 35: the higher the scores indicate higher addiction.
  For each of the three study arms, the change in total GAS scores between before the intervention and after the 12 week intervention is measured. Then, the average change scores in each of the three groups are compared with each other.

CONTACTS AND LOCATIONS:
Overall Officials: Hanna Renvall, PhD, Principal Investigator — Helsinki University Central Hospital
Locations (6):
- Finland (6):
  - Turku University Hospital, Turku, Southwest Finland
  - Aalto University (TMS), Espoo, Uusimaa
  - Aalto University, Department of Neuroscience and Biomedical Engineering, Espoo, Uusimaa
  - Helsinki University Hospital, Psychiatry, Helsinki, Uusimaa
  - Helsinki University Hospital BioMag laboratory, Helsinki, Uusimaa
  - University of Helsinki Neuroscience Center (MEG, MRI), Helsinki, Uusimaa

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lukka L, Vesterinen M, Salonen A, Bergman VR, Torkki P, Palva S, Palva JM. User journey method: a case study for improving digital intervention use measurement. BMC Health Serv Res. 2025 Apr 1;25(1):479. doi: 10.1186/s12913-025-12641-9. PMID 40165237